CLINICAL TRIAL: NCT06548555
Title: A Prospective Multicentric Study to Evaluate the Impact of Long-term Digital Education vs Standard of Care on LDL-C Levels in Post Myocardial Infarction Patients in the Czech Republic
Brief Title: A Study to Evaluate the Impact of Long-term Digital Education vs Standard of Care on LDL-C Levels in Post Myocardial Infarction Patients
Acronym: DEDUCA-CZ
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CKJX839A1CZ01
Record Dates: First submitted 2024-08-07; First posted 2024-08-12 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Myocardial Infarction
Keywords: myocardial infarction; MI; Czech Republic; secondary prevention; digital education; LDL-C
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Interventional arm: Patients receiving the systematic educational intervention
  Interventions: Other: systematic educational intervention
- Control arm: Patients treated in the clinical routine mode (the education of the patient follows routine practice and no added education is provided by the Healthcare Professionals).

INTERVENTIONS:
Other: systematic educational intervention — This is a non-interventional study and does not impose a therapy protocol, or a diagnostic/therapeutic procedure. Patients are treated according to the local prescribing information, and routine medical practice in terms of visit frequency and types of assessments performed and only these data is collected as part of the study.
  Groups: Interventional arm

SUMMARY:
The purpose of this study is to demonstrate the impact of digital education on the cardiovascular risk factors in post-Myocardial Infarction patients and to generate evidence for broad implementation of the proposed education program.

DETAILED DESCRIPTION:
The local (Czech Republic), multi-center, prospective, descriptive study, is a non-treatment interventional, two-armed stratified randomized (1:1), not blinded, controlled (parallel group) study in hospitalized adult patients after first myocardial infarction with two arms to evaluate the effect of systematic education program on the 12-months change of LDL-C. Patients are recruited (randomized) into two arms: interventional and control. The interventional arm receives the systematic educational intervention. The control arm is treated in the clinical routine mode, i.e., the education of the patient follows routine practice and no added education are provided by the HCPs (Healthcare Professionals). The post-MI treatment in both arms follows the standard of care (SOC). The End of Study (EOS) visit will be performed at month 12 at the place of the initial hospitalization.

The primary objective of the study is to describe the effect of the proposed educational program for post-MI patients on LDL-C at month 12 after the event compared to routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

Participants eligible for inclusion in this study must fulfil all the following criteria:

* Male or female patients ≥18 years of age,
* At the Screening Visit, participants must be hospitalized for the first myocardial infarction. This must be a spontaneous MI (either ST-elevation MI or non-ST-elevation MI), which was not the result of percutaneous coronary intervention (PCI) or coronary artery bypass graft (CABG). Confirmation of MI is a combination of signs or symptoms consistent with presentation of MI, and at least one of the following (adapted from (Thygesen, et al., 2018)):

  * Documentation of cardiac biomarkers that exceed the diagnostic threshold of a local laboratory for MI
  * Pathological Q waves on ECG or other ECG changes as defined in Appendix 2
  * Imaging evidence of loss of viable myocardium or regional wall motion abnormality in a pattern consistent with an infarction or ischemic etiology
  * Identification of a coronary thrombus by angiography at the time of presentation with MI,
* LDL-C ≥ 1.8 mmol/L at the time of the hospitalization,
* Ability to participate in the hybrid educational program (must be able to receive emails and watch online educational videos),
* Patients must provide written consent to participate in the study.

Exclusion Criteria:

Participants meeting any of the following criteria are not eligible for inclusion in this study:

* History of previous myocardial infarction,
* History of previous coronary intervention due to ASCVD (percutaneous coronary intervention (PCI) or coronary artery bypass graft (CABG)),
* History of ischemic stroke,
* Any surgical or medical condition, which in the opinion of the investigator, may place the participant at higher risk from his/her participation in the study, or is likely to prevent the participant from complying with the requirements of the study or completing the study,
* Patients diagnosed with homozygous familial hypercholesterolemia,
* Unwillingness or inability (e.g., physical, or cognitive) to comply with study procedures (including adherence to study visits and fasting blood draws) and schedule,
* Participation in any other interventional study, both treatment and non-treatment interventional study,
* Patients treated with inclisiran prior to the hospitalization for myocardial infarction.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients after the first myocardial infarction.
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2023-03-08 (Actual); Primary Completion 2024-10-24 (Actual); Study Completion 2024-10-24 (Actual)

PRIMARY OUTCOMES:
Absolute change in LDL-C levels from baseline at month 12 | Baseline, month 12
  Absolute change in LDL-C levels from baseline at month 12 after the event.
Relative (percentage) change in LDL-C levels from baseline at month 12 | Baseline, month 12
  Relative change in LDL-C levels from baseline at month 12 after the event.

SECONDARY OUTCOMES:
Percentage of patients achieving their LDL-C target level | Month 12
  Percentage of patients achieving their LDL-C target level according to the 2019 ESC/EAS Guidelines (LDL-C reduction of ≥50% from baseline and an LDL-C goal of <1.4 mmol/L)
Change in total cholesterol from Baseline at Month 12 | Baseline, month 12
  Change in total cholesterol from Baseline at Month 12
Change in HDL-C from Baseline at month 12 | Baseline, month 12
  Change in high-density lipoprotein cholesterol (HDL-C)
Change in VLDL-C from Baseline at month 12 | Baseline, month 12
  Change in very low- density lipoprotein cholesterol (VLDL-C).
Change in non-HDL-C from Baseline at month 12 | Baseline, month 12
  Change in non-high-density lipoprotein cholesterol (non-HDL-C).
Change in triglycerides from Baseline at month 12 | Baseline, month 12
  Change in triglycerides
Change in Lp(a) from Baseline at month 12 | Baseline, month 12
  Change in lipoprotein(a) [Lp(a)])
Blood pressure | Baseline, month 12
  Blood pressure at baseline and month 12 will be provided
Body Mass Index | Baseline, month 12
  BMI (Body Mass Index) at baseline and month 12 will be provided
Waist circumference | Baseline, month 12
  Waist circumference at baseline and month 12 will be provided
Number of patients smoking | Baseline, month 12
  Number of patients smoking at Baseline and at Month 12
Number of cigarettes smoked per week | Baseline, month 12
  Number of cigarettes smoked per week at Baseline and at Month 12
percentage of patients that have ceased smoking by Month 12 | Month 12
  percentage of patients that have ceased smoking by Month 12 after the event.
Percentage of patients that have changed their diet according to the recommendations | month 12
  Percentage of patients that have changed their diet according to the recommendations (such as increasing consumption of vegetables, fruits, whole grains, fish; reducing intake of trans-fats, sweets, sugar-added beverages and red meat) by Month 12 after the event.
Average number of units of alcohol consumed daily | Baseline, month 12
  Average number of units of alcohol consumed daily at Baseline and at Month 12
Percentage of patients that have decreased their alcohol intake | month 12
  Percentage of patients that have decreased their alcohol intake by Month 12 after the event.
Average estimated time spent by physical activities per week | Baseline, month 12
  Average estimated time spent by physical activities per week
Average number of steps walked daily | Baseline, month 12
  average number of steps walked daily at Baseline and Month 12.
Percentage of patients that have increased their physical activity | 12 months
  Percentage of patients that have increased their physical activity by Month 12 after the event.
Percentage of patients who registered at a cardiologist during the study | 12 months
  Percentage of patients who registered at a cardiologist during the study
Percentage of patients adherent to statin therapy | Baseline, month 12
  Percentage of patients adherent to statin therapy at baseline and at Month 12 in both arms. Adherence is defined as taking medications as prescribed >75% of the time based on responses to Gehi et al. adherence question ("In the past month, how often did you take statins as the doctor prescribed?") on Month 12
Number of participants by living conditions- family conditions | Baseline
  Living conditions- family conditions: marital status, number of children; place of residency (urban/rural)
Lipid profile | Baseline, month 12
  Lipid profile (LDL-C, total cholesterol, HDL-C, VLDL-C, non-HDL-C and triglycerides).
Lipid profile - Lp(a) | Baseline, month 12
  Lp(a) values at Baseline and month 12 will be provided
Number of participants with comorbidities | Baseline
  Comorbidities (diabetes mellitus, chronic kidney disease) at Baseline
Number of participants that manifest ASCVD in family history | Baseline
  Number of participants that manifest ASCVD in family history
Number of participants by MI pharmacological treatment | 12 months
  Number of participants by Myocardial Infarction (MI) pharmacological treatment
Percentage of patients treated with PCSK9 antibodies to patients eligible for PCSK9 antibodies | 12 months
  Percentage of patients treated with PCSK9 antibodies to patients eligible for PCSK9 antibodies (according to the Czech reimbursement criteria).

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- Czechia (4):
  - Novartis Investigative Site, Brno-Bohunice
  - Novartis Investigative Site, České Budějovice
  - Novartis Investigative Site, Ostrava Poruba
  - Novartis Investigative Site, Prague

IPD SHARING:
Plan to Share IPD: No